CLINICAL TRIAL: NCT02992652
Title: Role of Allopurinol in Prevention of Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Brief Title: Allopurinol in Prevention of Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 937
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): Received 600 mg of allopurinol divided in two oral doses before the procedure (300 mg at 15 hours and 300 mg at 3 hours before ERCP)
  Interventions: Drug: Allopurinol
- Control Group (No Intervention): Underwent ERCP without allopurinol prophylaxis

INTERVENTIONS:
Drug: Allopurinol — 600 mg of allopurinol divided in two oral doses before the procedure (300 mg at 15 hours and 300 mg at 3 hours before ERCP)
  Arms: Study Group

SUMMARY:
* The investigators evaluated the role of allopurinol in prevention of post-ERCP pancreatitis.
* 100 Egyptian patients who were candidates for ERCP were included and divided into two groups. Group 1 (study group) included 50 patients who received two doses of allopurinol 300 mg each, 15 hours and 3 hours before ERCP and Group 2 (control group) included 50 patients who did not receive allopurinol prophylaxis.

DETAILED DESCRIPTION:
A diagnosis of procedure-related pancreatitis was based on an increased serum amylase level greater than three times the upper normal limits, associated with abdominal pain requiring analgesics and persisting for at least 24 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were going to be subjected to ERCP due to different causes

Exclusion Criteria:

* Patients with clinically evident acute pancreatitis or hyperamylesemia (≥150 IU/L) before the procedure.
* Current or recent use of allopurinol (within the last 48 hours).
* Hypersensitivity to allopurinol or hydro-soluble contrast solutions.
* Current use of drugs with a known interaction with allopurinol, including cyclophosphamide, chlorpropamide, azathioprine, mercaptopurines, or probenecid.
* NSAIDS intake within a week prior to assessment.
* Previous endoscopic or surgical sphincterotomy.
* Those with severe co-morbid conditions.
* Female patients with a known or suspected pregnancy and/or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of procedure-related pancreatitis | At least 24 hours after the ERCP

IPD SHARING:
Plan to Share IPD: No